CLINICAL TRIAL: NCT05386277
Title: A Post Market Clinical Study to Confirm the Performance and Safety of the LeMaitre® TufTex Single Lumen Embolectomy Catheter on Patients Undergoing Surgical Treatment for the Removal of Arterial Emboli and/or Thrombi
Brief Title: A PMCF Study to Confirm the Performance and Safety of the LeMaitre® TufTex Single Lumen Embolectomy Catheter
Acronym: SLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LeMaitre Vascular (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC-16-001
Record Dates: First submitted 2022-05-10; First posted 2022-05-23 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Arterial Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LeMaitre TufTex Single Lumen Embolectomy Catheter (Other): The LeMaitre® Single Lumen Embolectomy Catheter is a catheter that consists of a natural latex rubber balloon secured with ligatures to a single lumen radiopaque shaft. When the balloon the emboli and/or thrombi can be removed by withdrawing the catheter tip through the arteriotomy.
  Interventions: Device: TufTex Single Lumen Embolectomy Catheter

INTERVENTIONS:
Device: TufTex Single Lumen Embolectomy Catheter — The SLC Embolectomy Catheter is indicated for the removal of arterial emboli and thrombi

SUMMARY:
A post market clinical study to confirm the performance and safety of the LeMaitre® TufTex Single Lumen Embolectomy Catheter on patients undergoing surgical treatment for the removal of arterial emboli and/or thrombi

DETAILED DESCRIPTION:
This prospective, single arm, post market clinical study was designed to proactively collect clinical data on the LeMaitre® TufTex Single Lumen Embolectomy Catheters and to confirm its performance in removing arterial emboli and/or thrombi, to identify and analyze emergent risks on the basis of factual evidence, and to ensure the continued acceptability of the benefit/risk ratio. This post market study is sponsored by LeMaitre® Vascular, Inc., the manufacturer of the device. Study will take place at 3 to 8 sites in Europe, the target sample size is 112 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subject, ≥ 18 years of age at time of enrollment.
2. Subject who is scheduled to undergo surgical treatment for the removal of arterial or venous emboli and/or thrombi, where one of the LeMaitre® Embolectomy Catheter will be used.
3. Subject signed an Informed Consent for participation.
4. Subject diagnosed with a embolus/thrombus.
5. Subjects for whom thrombolytic therapy had failed or was contraindicated.

Exclusion Criteria:

1. Co-morbidity that in the discretion of the investigator might confound the results.
2. Subjects who are unable to read or write.
3. Pregnant or lactating women at time of enrollment
4. Subjects who are immune comprised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety objective is defined as acceptable safety outcomes (e.g. (Serious) Device and/or Procedure Related Events) during the procedure | During procedure and 1 month post index procedure
  The primary safety objective is defined as acceptable safety outcomes (e.g. (Serious) Device and/or Procedure Related Events) during the procedure and 1 Month post index procedure.
Performance objective is the technical success as defined as <30% residual stenosis | 1 month post index procedure
  The primary performance objective is the technical success as defined as <30% residual stenosis of the target vessel.

SECONDARY OUTCOMES:
1. Clinical success | 1 Month after the index procedure
  Clinical success is target vessel dependent and defined as; (1) The absence of target vessel limb amputation post-intervention in case of limb cloths, and 2. successful dialysis sessions performed post-intervention in case of dialysis shunt revascularization (2) Revision rate is defined as the number of patients with target vessel reintervention (3) Primary assisted patency is defined as target vessel patency; the target vessel is patent but there may have been some intervention required to maintain that patency. (4) Secondary patency is defined as the target vessel patency including target vessel that have been occluded and there has been an intervention to restore patency.
2. Revision Rate | 1 month post index procedure
  Revision rate is defined as the number of patients with target vessel reintervention
3. Primary Assisted Patency | 1 month post index procedure
  Primary assisted patency is defined as target vessel patency; the target vessel is patent but there may have been some intervention required to maintain that patency.
4. Secondary Patency | 1 month post index procedure
  Secondary patency is defined as the target vessel patency including target vessel that have been occluded and there has been an intervention to restore patency.

OTHER OUTCOMES:
Exploratory endpoints | 1 month post index procedure
  Number of LeMaitre® Embolectomy Catheters used per intervention Number of balloon tears per intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Prouse, Principal Investigator — Ospedale Regionale di Lugano - sede Civico
Locations (3):
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Andrej Udelnow, Brandenburg, Germany
- Giorgio Prouse, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No